CLINICAL TRIAL: NCT00964249
Title: Phase I Study of GW642444M- A Randomized, Double Blind, Placebo Controlled, Parallel-group, 7 Day Repeat Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Inhaled Dose of GW642444M From a Novel Dry Powder Device in Healthy Japanese Male Subjects -
Brief Title: Phase I Study of GW642444M in Healthy Japanese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 112017; NCT00753701 (obsolete NCT alias)
Record Dates: First submitted 2009-08-13; First posted 2009-08-24 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- LABA (Experimental): After randomization subject will inhale either 12.5 microgram or 25 microgram GW642444M once daily for 7 days.
  Interventions: Drug: GW642444
- Placebo (Placebo Comparator): After randomization subjects will inhale placebo once daily for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GW642444 — Long acting Beta 2 agonist
  Arms: LABA
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double blind, placebo controlled, parallel-group, 7 day repeat dose study to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of inhaled dose of GW642444M from a novel dry powder device in healthy Japanese male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Japanese healthy male subjects aged between 20 and 64 years of age inclusive. Healthy subjects are defined as individuals who are free from clinically significant illness or disease as determined by their medical history, physical examination, laboratory studies, and other tests.
2. Body weight ≥ 50kg and BMI within the range 18.5-25.0kg/m2 inclusive.
3. Non-smokers (never smoked or not smoking for >6 months with <10 pack years history (Pack years = (cigarettes per day smoked/20) x number of years smoked))
4. Normal spirometry (FEV1 ≥ 80% of predicted, FEV1/FVC ≥ 70%).
5. Clinical laboratory tests data obtained at screening meet the following:

   AST(GOT), ALT(GPT), total-bilirubin: below the upper limit of the normal ranges
6. Serum potassium and glucose within normal range at screening
7. Normal 12-lead EGC finding at screening; QTc interval <450msec
8. A mean heart rate within the range 40-90 beats per minute (bpm) inclusive at screening.
9. A mean blood pressure lower than 140/90mmHg at screening.
10. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
11. Capable of using the novel dry powder inhaler.

Exclusion Criteria:

1. The subject has any clinically relevant abnormality on medical examination, vital sign, clinical laboratory test or medical history at screening in the medical opinion of the investigator or the subject has a medical history that is not considered as eligible for inclusion in this study by the investigator.
2. The subject is currently participating in another clinical study or post-marketing study in which the subject is or will be exposed to an investigational or a non-investigational drug or device.
3. The subject has participated in a clinical study with an investigational or a non-investigational drug or device during the previous 4 months.
4. A history of breathing problems (i.e. history of asthmatic symptomatology, asthma in childhood).
5. The subject has an allergy for any drug or idiosyncrasy
6. The subject has a known allergy or hypersensitivity to milk protein or the excipients lactose monohydrate and magnesium stearate.
7. The subject has a history or current conditions of drug abuse or alcoholism.
8. History of regular alcohol consumption exceeding on average, 14 drinks/week (1 drink=5 ounces (150mL) of wine or 350mL of beer or 1.5 ounces (45mL) of 80 proof distilled spirits) within 6 month of screening.
9. The subject is positive for urine drug screening.
10. Use of prescription or non-prescription drugs, including CYP3A/PGP inhibitor, vitamins, herbal and dietary supplements (including St John'sWort) within 14 days prior to the first dose of study medication.
11. The subject is positive for syphilis, HBs antigen, HCV antibody, HIV antibody, HTLV-1 antibody.
12. The subject has donated a unit of blood ">400mL" within the previous 4 months or ">200mL" within the previous 1 month.

Ages: 20 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-09-20 (Actual); Primary Completion 2008-12-01 (Actual); Study Completion 2008-12-01 (Actual)

PRIMARY OUTCOMES:
Safety：adverse events, vital sign, ECGs, and clinical laboratory test
PK：Cmax, tmax and AUC(0-t)

SECONDARY OUTCOMES:
Pharmacodynamics parameters of the systemic β-adrenergic effect (heart rate, blood pressure, QTc, glucose and potassium)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Nakahara N, Wakamatsu A, Kempsford R, Allen A, Yamada M, Nohda S, Hirama T. The safety, pharmacokinetics and pharmacodynamics of a combination of fluticasone furoate and vilanterol in healthy Japanese subjects. Int J Clin Pharmacol Ther. 2013 Aug;51(8):660-71. doi: 10.5414/CP201822. PMID 23735179
- See also: Results for study 112017 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/112017?search=study&search_terms=112017#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 112017 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112017 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112017 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112017 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112017 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register